CLINICAL TRIAL: NCT05434234
Title: A Phase 1A/1B, Multicenter, Nonrandomized, Open-Label, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of YL201 as a Single Agent and in Combination With Other Anti-Cancer Therapies in Patients With Advanced Solid Tumors
Brief Title: A Study of YL201 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YL201-INT-101-01
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
Keywords: Antibody-drug conjugate
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation (Experimental): All participants enrolled in the dose escalation part
  Interventions: Drug: YL201
- Dose expansion (Experimental): All participants enrolled in the dose expansion part
  Interventions: Drug: YL201
- Dose Selection (Experimental)
  Interventions: Drug: YL201 and atezolizumab

INTERVENTIONS:
Drug: YL201 — Patients will be treated with YL201 intravenous (IV) infusion once every 3 weeks (Q3W) as a cycle.
  Arms: Dose escalation
Drug: YL201 — Patients will be treated with YL201 intravenous (IV) (A mg/kg or B g/kg infusion once every 3 weeks (Q3W) as a cycle.
  Arms: Dose expansion
Drug: YL201 and atezolizumab — Patients will be treated with YL201 intravenous (IV) infusion (A mg/kg or B mg/kg, up to 200mg) followed by atezolizumab on day 1 of each 21 day cycle
  Arms: Dose Selection

SUMMARY:
This is a phase 1, multicenter, nonrandomized, open-label, first-in-human study of YL201 conducted in China and the United States. The study will include 2 parts: a dose escalation part (Part 1) followed by a dose expansion part (Part 2).

Part 1 will estimate the MTD/RED(s) in dose escalation cohorts of patients with advanced solid tumors unresponsive to currently available therapies or for whom no standard therapy is available.

Part 2 will include patients with selected advanced solid tumor types enrolled at the MTD/RED(s), to better define the safety profile and evaluate the efficacy of YL201.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the trial before the start of the trial and voluntarily sign their name and date on the ICF
* Aged ≥18 years
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Adequate organ and bone marrow function
* Female patients of childbearing potential must agree to use a highly effective form of contraception and not donate, or retrieve for their own use, ova from the time of screening and throughout the study period, and for at least 5 months after the last dose of atezolizumab or 6 months after the last dose of YL201, whichever is later. Male patients must agree to use a highly effective form of contraception and not freeze or donate sperm from the time of screening and throughout the study period, and for at least 6 months after the last dose of YL201.
* Life expectancy of ≥3 months
* Able and willing to comply with protocol visits and procedures
* Have at least 1 evaluable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Pathologically confirmed diagnosis of an advanced solid tumor (SCLC, mCRPC, ESCC and NSCLC are preferred) for which standard treatment had proven to be ineffective or intolerable, or no standard treatment is available. For ES-SCLC patients in Arm C: no prior anti-cancer treatment

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study
* Prior systemic anticancer treatment including chemotherapy, molecular -targeted therapy, hormonal therapy, immunotherapy, or biological therapy within 3 weeks before the first dose of study drug (use of oral fluorouracil [eg, tegafur and capecitabine] or small molecular-targeted therapy within 2 weeks or 5 half-life periods [whichever is shorter]before the first dose; use of mitomycin or nitrosoureas within 6 weeks before the first dose; use of herbal medicine with antitumor indications or nonspecific immunomodulators [eg, thymosin, interferon, and interleukin] within 2 weeks before the first dose).
* Prior radiation therapy, including palliative stereotactic radiation with abdominal, within 4 weeks before the first dose of study drug (if palliative stereotactic radiation therapy without abdominal, within 2 weeks)
* Undergone major surgery (not including diagnostic surgery) within 4 weeks before the first dose of study drug or expect major surgery during the study
* Undergone allogeneic hematopoietic stem cell transplantation (HSCT) before the first dose of study drug, or autologous HSCT within 3 months before the first dose of study drug
* Received systemic steroids (>10 mg/day of prednisone or its equivalent) or other immunosuppressive therapy within 2 weeks before the first dose of study drug. Received any live vaccine within 4 weeks before the first dose of study drug or intend to receive a live vaccine during the study
* Known human immunodeficiency virus (HIV) infection
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Active HBV is defined as hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) positive, and HBV DNA level above ULN at the study site; active HCV is defined as positive hepatitis C antibody and HCV RNA level above ULN at the study site
* Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia and pigmentation) not yet resolved to NCI CTCAE Grade ≤1, baseline, or the level specified in the inclusion/exclusion criteria. Patients with chronic Grade 2 toxicities who are asymptomatic or adequately managed with stable medication may be enrolled after discussion with the sponsor
* A history of severe hypersensitivity reactions to the drug substances, inactive ingredients in the drug product, or other mAbs
* Women who are breastfeeding or pregnant as confirmed by pregnancy tests performed within 7 days before the first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2027-04-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the occurrence of DLTs during the first cycle in Part 1 | 21 days of Cycle 1
Evaluate the AEs in Part 2 as characterized by type, frequency, severity, timing, seriousness and relationship to study treatment | By the global end of trial date, approximately within 36 months
Evaluate the prostate-specific antigen (PSA) response rate for patients with prostate cancer in Part 2 | Approximately within 36 months
  PSA response rate: defined as the proportion of patients who achieved a ≥50% decrease in PSA from baseline
Evaluate the objective response rate (ORR) for patients with solid tumors other than prostate cancer in Part 2, assessed using RECIST version 1.1 | Approximately within 36 months
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).
Laboratory abnormalities as characterized by type, frequency, severity, and timing in Part 2 | Biy the end of trial date, approximately within 36 months
Incidence, nature, and severity of AEs graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V5.0 in Part 3 | Biy the end of trial date, approximately within 36 months
Nature and frequency of dose-limiting toxicities (DLTs), incidence, nature, and severity of laboratory abnormalities in Part 3 | At the end of cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
Evaluate the AEs in Part 1 as characterized by type, frequency, severity, timing, seriousness and relationship to study treatment | By the global end of trial date, approximately within 36 months
Characterize the PK parameter AUC | Approximately within 36 months
Characterize the PK parameter Cmax | Approximately within 36 months
Characterize the PK parameter Ctrough | Approximately within 36 months
Characterize the PK parameter CL | Approximately within 36 months
Characterize the PK parameter Vd | Approximately within 36 months
Characterize the PK parameter t1/2 | Approximately within 36 months
Assess the incidence of anti-YL201 antibodies | Approximately within 36 months
Evaluate the prostate-specific antigen (PSA) response rate for patients with prostate cancer in Part 1 | Approximately within 36 months
  PSA response rate: defined as the proportion of patients who achieved a ≥50% decrease in PSA from baseline
Evaluate the PSA progression-free survival (PSA-PFS) for patients with prostate cancer | Approximately within 36 months
  PSA-PFS: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of PSA progression, based on PCWG3 criteria.
Evaluate the radiological PFS (rPFS) for patients with prostate cancer | Approximately within 36 months
  rPFS: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of radiographic tumor progression or death due to any cause, whichever occurs first, based on RECIST 1.1 and PCWG3 criteria.
Evaluate the failure-free survival (FFS) for patients with prostate cancer | Approximately within 36 months
  FFS: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of radiographic tumor progression, unequivocal clinical progression, PSA progression or death due to disease progression, whichever occurs first.
Evaluate the objective response rate (ORR) for patients with solid tumors other than prostate cancer in Part 1, Part 2, and Part 3, assessed using RECIST version 1.1 | Approximately within 36 months
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).
Evaluate the disease control rate (DCR) for patients with solid tumors other than prostate cancer, assessed using RECIST version 1.1 | Approximately within 36 months
  DCR: defined as the proportion of patients who achieved a best overall response of CR, PR or stable disease (SD).
Evaluate the duration of response (DoR) for patients with solid tumors other than prostate cancer, assessed using RECIST version 1.1 | Approximately within 36 months
  DoR: defined as the time interval from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of PD. DoR will be assessed for patients with a response (CR or PR) only.
Evaluate the time to response (TTR) for patients with solid tumors other than prostate cancer, assessed using RECIST version 1.1 | Approximately within 36 months
  TTR: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of objective response (CR or PR).
Evaluate the progression-free survival (PFS) for patients with solid tumors other than prostate cancer, assessed using RECIST version 1.1 | Approximately within 36 months
  PFS: defined as the time interval from the date of the first dose of study drug to the date of first documentation of PD or death due to any cause, whichever occurs first.
Evaluate the overall survival (OS) for patients with solid tumors | Approximately within 36 months
  OS: defined as the time interval from the date of the first dose of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (19):
  - 002, Fair Oaks, California
  - 001, La Jolla, California
  - 003, Lone Tree, Colorado
  - 004, Washington D.C., District of Columbia
  - 005, Boston, Massachusetts
  - 006, Ann Arbor, Michigan
  - 007, Detroit, Michigan
  - 008, St Louis, Missouri
  - 009, Santa Fe, New Mexico
  - 010, New York, New York
  - 011, Chapel Hill, North Carolina
  - 012, Nashville, Tennessee
  - 014, Houston, Texas
  - 015, Irving, Texas
  - 013, San Antonio, Texas
  - 016, Tyler, Texas
  - 017, Fairfax, Virginia
  - 018, Spokane, Washington
  - 019, Tacoma, Washington
- Canada (4):
  - 020, Edmonton, Alberta
  - 021, Kelowna, British Columbia
  - 022, Brampton, Ontario
  - 023, Toronto, Ontario
- China (2):
  - 024, Guangzhou, Guangdong
  - 025, Zhengzhou, Henan
- France (8):
  - 026, Bordeaux
  - 027, Dijon
  - 028, Marseille
  - 029, Nantes
  - 030, Paris
  - 031, Poitiers
  - 032, Saint-Herblain
  - 033, Suresnes
- Poland (2):
  - 044, Otwock
  - 045, Poznan
- Spain (10):
  - 034, Barcelona, Barcelona
  - 035, Barcelona, Barcelona
  - 039, Leganés, Madrid
  - 037, Madrid, Madrid
  - 036, Madrid, Madrid
  - 038, Moncloa-Aravaca, Madrid
  - 041, Pozuelo de Alarcón, Madrid
  - 042, Usera, Madrid
  - 040, Pamplona, Navarre
  - 043, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma Y, Yang Y, Huang Y, Fang W, Xue J, Meng X, Fan Y, Fu S, Wu L, Zheng Y, Liu J, Liu Z, Zhuang W, Rosen S, Qu S, Li B, Li M, Zhao Y, Yang S, Ji Y, Sommerhalder D, Luo S, Yang K, Li J, Lv D, Zhang P, Zhao Y, Hong S, Zhang Y, Zhao S, Chin S, Zhang X, Lian W, Cai J, Xue T, Zhang L, Zhao H. A B7H3-targeting antibody-drug conjugate in advanced solid tumors: a phase 1/1b trial. Nat Med. 2025 Jun;31(6):1949-1957. doi: 10.1038/s41591-025-03600-2. Epub 2025 Mar 13. PMID 40082695